CLINICAL TRIAL: NCT05477290
Title: A Comparative Study of Hand Function and Scar-Related Health-Related Quality of Life in Trigger Finger Release
Brief Title: Function and Scar in Trigger Finger Release
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Achilleas Thoma, Surgeon, McMaster University
Other Study IDs: 7242
Record Dates: First submitted 2022-07-13; First posted 2022-07-28 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Trigger Finger
Keywords: Scar; Function; Health-Related Quality of Life
MeSH Terms: conditions — Trigger Finger Disorder; Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Transverse incision: At the level of the A1 pulley, a transverse incision will be made and the flexor pulley will be exposed with blunt dissection. The pulley will be transected and the wound will subsequently be closed with 4.0 Monocryl after ensuring complete release
  Interventions: Procedure: Trigger Finger Release through Transverse Incision
- Oblique incision: At the level of the A1 pulley, a oblique incision will be made and the flexor pulley will be exposed with blunt dissection. The pulley will be transected and the wound will subsequently be closed with 4.0 Monocryl after ensuring complete release.
  Interventions: Procedure: Trigger Finger Release through Oblique Incision
- Vertical incision: At the level of the A1 pulley, a vertical incision will be made and the flexor pulley will be exposed with blunt dissection. The pulley will be transected and the wound will subsequently be closed with 4.0 Monocryl after ensuring complete release.
  Interventions: Procedure: Trigger Finger Release through Vertical Incision

INTERVENTIONS:
Procedure: Trigger Finger Release through Transverse Incision — At the level of the A1 pulley, a transverse incision will be made and the flexor pulley will be exposed with blunt dissection. The pulley will be transected and the wound will subsequently be closed with 4.0 Monocryl after ensuring complete release.
  Groups: Transverse incision
Procedure: Trigger Finger Release through Oblique Incision — At the level of the A1 pulley, a oblique incision will be made and the flexor pulley will be exposed with blunt dissection. The pulley will be transected and the wound will subsequently be closed with 4.0 Monocryl after ensuring complete release.
  Groups: Oblique incision
Procedure: Trigger Finger Release through Vertical Incision — At the level of the A1 pulley, a vertical incision will be made and the flexor pulley will be exposed with blunt dissection. The pulley will be transected and the wound will subsequently be closed with 4.0 Monocryl after ensuring complete release.
  Groups: Vertical incision

SUMMARY:
Trigger finger is a common upper limb impairment associated with a significant decrease in quality of life, hand dexterity and strength as well as increased pain while complying daily activities of living. Trigger finger can be managed through the surgical release of the ligaments in the affected finger. The open surgical release of trigger finger can be accomplished through multiple incision types. As such, each incision may present different risks of harming or disturbing the underlying anatomy in the hand. This study aims to assess the variation in three incisional techniques (oblique, transverse and vertical) to determine which incision is preferential to improve scar aesthetics, increase hand function and minimize complications. Patients will be observed following surgery and information about hand function and quality of life will be obtained through the administration of questionnaires. Data will be collected at four time-points, one prior to and three following surgery.

DETAILED DESCRIPTION:
A study describing the superior incision technique is still needed to assess post-open release outcomes of the surgical site such as aesthetics and hand function. This study contributes to literature by providing further clarification into which technique of open trigger finger release is preferential to optimize scar aesthetics, increase function and, minimize complications using patient reported outcome measures such as the MHQ and SCAR-Q. The primary objective of this study is to assess patient Health-Related Quality of Life related to hand function via three incisional techniques using the generic hand instrument, (MHQ). This will be measured at 1 week prior, 1 day prior, and 1, 3, and 6 months post operation. The secondary objective will be to evaluate the Health-Related Quality of Life related to scar appearance post trigger finger release of three (transverse, oblique and vertical) incisional techniques of trigger finger release using the SCAR-Q (a condition-specific scales) at 1, 3 and 6 months post operation.

This study will be employed as a three-arm prospective cohort study. Local surgeons practicing at St. Joseph's Healthcare who utilize different incisional techniques for trigger finger release will compare each of their techniques. As each group sees trigger finger at a roughly equal rate, it is expected that the target of 30 patients in each group will be met in a similar timeline. Data will be recorded by a research team member that is not the operating physician via a paper-based system specific to this study.

At consultation patients will be approached for consent within a private consultation room within the surgical clinic. One week prior to surgery patients will complete questionnaires at the principle investigator's office (completed by the RA) in a private room. Post operation, patients will return to the principle investigator's office at 1, 3, 6 and 12 months post operation to complete the same questionnaires and to document any complications they have experienced.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Trigger finger release of the 2nd, 3rd, 4th, or 5th finger
* Diagnosed stenosing tenosynovitis or trigger finger prior to release
* Able to understand and communicate English

Exclusion Criteria:

1. Previous attempted surgical treatment
2. Patients undergoing any concomitant procedure on the same hand (e.g. carpal tunnel release)
3. Patients who are unable to provide informed consent.
4. Patients who do not have a fixed address

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals receiving trigger finger release surgery from surgeons who are co-investigators in this study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life related to hand function | 1 week prior, 1 day prior, and 1, 3 and 12 months post operation
  Outcome measured through the Michigan Hand Questionnaire (MHQ). The MHQ has a total score of 100; the lowest possible score is 0. A score of 100 on the MHQ indicates the best possible ability.

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life related to scar appearance | 1 week prior, 1 day prior, and 1, 3 and 12 months post operation
  Scar appearance, symptoms and the psychosocial impact of the scar will be measured using the SCAR-Q. This questionnaire has a minimum score of 0 and a maximum score of 100 with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Achilles Thoma, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
we do not plan on sharing data with other researchers